CLINICAL TRIAL: NCT02014532
Title: The Effect Of SRP With Adjunctive Systemic Therapy Of Leukotriene Receptor Antagonist-Montelukast On The Serum C Reactive Protein Levels & Clinical Parameters In Chronic Periodontitis Patients - A Randomized Controlled Trial
Brief Title: Role of Leukotriene Receptor Antagonists in Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr.Saurabh Inamdar, Principal Investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TKDC15
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Periodontitis
Keywords: Leukotriene receptor antagonist; Chronic periodontitis; Scaling and root planing; C- reactive protein
MeSH Terms: conditions — Chronic Periodontitis | interventions — montelukast; Leukotriene Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast (Active Comparator): Patients in Test Group were given Leukotriene receptor antagonist, Montelukast 1 tablet twice daily for 3 weeks then medications were stopped and changes in all parameters were again checked after 6 weeks.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Patients in Control Group were given placebo drug 1 tablet twice daily for 3 weeks then medications were stopped and changes in all parameters were again checked after 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Patients in Montelukast Group were treated with scaling and root planing (SRP) along with Montelukast (Montair 10mg), 1 tablet twice daily for 3 weeks.
  Other Names: Montair 10 mg (brand name); Leukotriene receptor antagonist.
  Arms: Montelukast
Drug: Placebo — Patients in Placebo Group were treated with scaling and root planing (SRP) along with Placebo therapy, 1 tablet twice daily for 3 weeks.
  Arms: Placebo

SUMMARY:
The adjunctive use of Leukotriene Receptor Antagonist (Montelukast) along with scaling and root planing in patients with chronic periodontitis leads to host inflammatory response modulation and decrease in serum C reactive protein (CRP) levels. If proven this will open new vistas in treatment of chronic periodontitis.

DETAILED DESCRIPTION:
A RCT was carried out to check the efficacy of Montelukast as an adjunct to scaling and root planing. The patients were randomised to either test group (SRP + Montelukast) and control group (SRP). Clinical parameters were assessed at baseline, 3 weeks and 6 weeks. Serum C-reactive protein levels were assessed at baseline, 3 weeks and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients within age group of 30 to 55 years.
2. Systemically healthy individuals.
3. Patients with chronic generalized periodontitis (moderate and severe) according to Center of Disease Control (CDC) working group, 2007 criteria

Exclusion Criteria:

1. Patients with systemic illnesses (i.e., diabetes mellitus, cancer, human immunodeficiency syndrome, bone metabolic diseases, or disorders that compromise wound healing, radiation, or immunosuppressive therapy),
2. Smoking,
3. Chronic alcoholics,
4. Pregnancy or lactation,
5. Use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), steroids or antibiotics / antimicrobials within January 2012 to Jun 2013,
6. Confirmed or suspected intolerance to Montelukast,
7. Periodontal therapy done within the January 2012 to Jun 2013.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the serum C- reactive protein levels at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  The biochemical parameter of serum C- reactive protein levels were checked at baseline, 3 weeks and 6 weeks. Montelukast therapy was started at baseline and continued for 3 weeks in test group and the post treatment levels were further checked at 6 weeks (i.e. 3 weeks after stoppage of Montelukast.) the change in C- reactive protein levels was analysed.
Changes from baseline in the probing pocket depth at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks.
  The probing pocket depths were checked at baseline, 3 weeks and 6 weeks. Montelukast therapy was started at baseline and continued for 3 weeks in test group and the post treatment levels were further checked at 6 weeks (i.e. 3 weeks after stoppage of Montelukast.) The change in probing pocket depth was analysed.
Changes from baseline in the clinical attachment level at 3 weeks and 6 weeks. | baseline, 3 weeks and 6 weeks
  The clinical attachment levels were checked at baseline, 3 weeks and 6 weeks. Montelukast therapy was started at baseline and continued for 3 weeks in test group and the post treatment levels were further checked at 6 weeks (i.e. 3 weeks after stoppage of Montelukast.) The change in clinical attachment levels was analysed.

SECONDARY OUTCOMES:
Changes from baseline in Gingival Index (GI) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, GI were assessed at 3 weeks after starting therapy with Montelukast, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. GI has a scoring criteria specified by Silness & Loe, 1963.
Changes from baseline in Plaque Index (PI) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, PI were assessed at 3 weeks after starting therapy with Montelukast, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. PI has a scoring criteria specified by Loe & Silness, 1964.
Changes from baseline in Oral Hygiene Index-Simplified (OHI-S) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, OHI-S were assessed at 3 weeks after starting therapy with Montelukast, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. OHI-S has a scoring criteria specified by Greene and Vermilion, 1964.
Changes from baseline in Sulcus Bleeding Index (SBI) at 3 weeks and 6 weeks | baseline, 3 weeks and 6 weeks
  changes from baseline in standard clinical parameter, SBI were assessed at 3 weeks after starting therapy with Montelukast, then therapy was stopped and same changes were again assessed at 6 weeks from baseline. SBI has a scoring criteria specified by Muhleman (1971).

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh P Inamdar, BDS, Principal Investigator — Post Graduate student
Locations (1):
- Tatyasaheb Kore Dental College and Research Centre, New Pargaon, Kolhāpur, Maharashtra, India